CLINICAL TRIAL: NCT02789722
Title: Application of Yerba Mate (Ilex Paraguariensis A.St.-Hil.) Products on the Promotion of Health: Assessment of Cardiovascular Health
Brief Title: Yerba Mate (Ilex Paraguariensis A.St.-Hil.): Assessment of Cardiovascular Health
Acronym: YMCH-2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karimi Sater Gebara (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor-Investigator, Karimi Sater Gebara, Master, Universidade Paranaense
Organization: Universidade Paranaense (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UNP-ILCV-1518
Record Dates: First submitted 2016-02-28; First posted 2016-06-03 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Disease; Diabetes
Keywords: Mate; Vascular protection; Endothelial function; Ilex paraguariensis
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yerba Mate Extract 750 mg (Experimental): Yerba Mate Extract - Capsules: daily dose of 2.250 g, distributed in 3 doses of 750 mg, for 28 days.
  Interventions: Other: Yerba Mate Extract
- Placebo (Placebo Comparator): Starch - Capsules: 3 times daily for 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Yerba Mate Extract — Yerba Mate extract capsules 750 mg
  Arms: Yerba Mate Extract 750 mg
Other: Placebo — Take 3 capsules, 3 times daily for 28 days.
  Arms: Placebo

SUMMARY:
Mate or yerba-mate (Ilex paraguariensis A.St.-Hil.) is a native plant from South America highly consumed in this region. Different traditional products (mate, mate tea, chimarrao, tereré) are obtained from the yerba-mate leaves and consumed as herbal tea. Mate is a rich source of bioactive phenolic compounds, mainly caffeoylquinic acids. The richness of different mono- and dicaffeoylquinic acids is a peculiarity of mate derived products. However, in contrast to other plant-based beverages rich in polyphenols like tea or coffee, the research and the industry have yet little explored the potential interest of mate product to promote human health. There has been a growing interest to the development of healthier foods to face the burden of cardiovascular diseases (CVD), especially those naturally rich in bioactive phenolic compounds with protective effects against the development of chronic diseases. Different in vitro and animals studies associate the mate consumption with cardiovascular protection mechanisms. Consistent information about this activity and the long-term consumption effects in humans are scarce. The aim of this study is to assess through a randomized controlled trial the impact of chronic intake of mate on intermediate biomarkers of cardiovascular health in humans and to identify possible involved nutrigenomic mechanisms.

DETAILED DESCRIPTION:
Mate is a traditional drink obtained from the leaves of yerba-mate (Ilex paraguariensis A.St.-Hil.), a native species of South America that has a great regional importance. Mate is highly consumed in South America countries because of the tradition acquired from the native populations. In these countries, mate is consumed as largely as tea (camellia sinensis) in Asia and Europe and coffee in Europe and North America. Mate constitutes a raw material little explored compared to other plant products like coffee or tea. However, mate product has recently raised interest due to both its high content of phytochemicals and the peculiarity of its phenolic profile, characterized by the wealth in mono and dicaffeoylquinic acids, known for their biological activities.

A large number of in vitro studies have evaluated the antioxidant capacity of mate products with different methodologies, and showed that the antioxidant effect was related to the presence of caffeoyl derivatives. Mate appears as a potent inhibitor of low-density lipoproteins (LDL) oxidation. The phenolic compounds of mate also exhibit free radical scavenging properties and inhibit a chemically induced oxidation of lipid in membranes. Different animal studies have reported a positive impact of mate consumption on some cardiovascular risk factors. These published data, obtained in different rodent models of diet induced dyslipidemia, obesity or atherosclerosis, suggest that the supplementation with mate products may improve plasma lipids profile, prevent hepatic fatty deposition, reduce insulin resistance, improve endothelial function and inhibit atherosclerosis progression. Few clinical studies reported positive effects of mate consumption on the blood lipid profile, glycemia and anthropometric parameters in healthy and unhealthy subjects.

The aim of this study is to assess through a randomized controlled trial the impact of chronic intake of mate on intermediate biomarkers of cardiovascular health in humans and to identify possible nutrigenomic mechanisms involved.

The study consists in a controlled, randomized, double blind, crossover clinical trial. This study will involve 36 healthy middle-age (45-65) male subjects selected according to the inclusion and exclusion criteria previously established. The study will have a maximum duration of 84 days including the wash-out period. The volunteers will have to consume daily for 4 weeks the mate extract (with a standardized content in phenolic compounds) or the placebo. At the beginning and/or at the end of each experimental period, blood will be sampled for measurement of glycemic and lipidic parameters, inflammatory markers and transcriptome analysis. Urine samples will also be collected for metabolomics analysis to characterize the exposure profile of volunteers in response to mate phenolic compounds consumption.

ELIGIBILITY:
Inclusion Criteria:

* No smoking, or having stopped smoking for more than three years;
* Having no more than one of the five criteria associated with metabolic syndrome proposed by the National Cholesterol Education Program's Adult Treatment Panel III (NCEP-ATP III) and approved by Brazilian scientific societies in the First Brazilian Guideline for Diagnosis and Treatment of Metabolic Syndrome (2005);
* Not consuming multivitamin supplements, antioxidants or polyphenols rich products in the last 3 months before the study;
* Accepting reduced consumption of natural polyphenols rich beverages (yerba mate, tea, coffee, wine, cocoa, soy milk, fruit juices) during the study;
* Not using any antihypertensive or anticholesterolemic drugs;
* Accepting to participate in the study after signing the Informed Consent and completing the information document.

Exclusion Criteria:

* Being diagnosed with diabetes, mental illness or other severe conditions that may influence the results of the study;
* Chronic alcoholism;
* Having severe hypertension with clinical complications such as acute myocardial infarction and other coronary artery diseases;
* Having kidney or liver diseases;
* Not accepting to participate in the study refusing to sign the Informed Consent, in accordance with the fundamental ethical and scientific requirements.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Quantification of biochemical parameters: total cholesterol and fractions, triglycerides and fasting glucose. | 28 days
  Cholesterol - Enzymatic colorimetric method; HDL cholesterol - lipoproteins VLDL (very low density lipoprotein) and LDL (Low Density Lipoprotein) and chylomicrons are precipitated with a mixture of phosphotungstic acid and magnesium chloride. After centrifugation, the bound cholesterol to high density lipoproteins (HDL) in the supernatant determined by colorimetric enzymatic method; Triglycerides - Enzymatic colorimetric method; Fasting glucose - enzymatic colorimetric method.
  All results are expressed in mg / dL.
Quantification of inflammatory markers: C-reactive protein. | after 28 days of treatment
  C-reactive protein (CRP) - Kit using turbidimetric methods for the quantitative
Quantification of adhesion molecule:Endothelin, Intercellular adhesion molecule (ICAM-1) and vascular endothelial cell adhesion molecule (VCAM-1). | 28 days
  Endothelin (EDN-1) - using enzyme immunoassay kit (ELISA) for the quantification in vitro EDN-1 in human serum. Evaluation kit for using enzyme immunoassay technique (ELISA) for the quantitative in vitro determination of ICAM-1 and VCAM-1 in human serum. The results of analyzes are expressed in ng/ml.
Quantification of inflammatory markers: Interleukin-6. | after 28 days of treatment
  Interleukin-6 (IL-6) - Evaluation kit for using enzyme immunoassay technique (ELISA) for the quantitative determination of IL-6 in vitro in human serum. The results of analyzes for IL-6 are expressed in ng/ml.
Evaluation of the tolerance glucose. | after 28 days of treatment
  Oral Glucose Tolerance Test OGTT (in mg/dL). A standard anhydrous glucose load will be administered and evaluation of Oral Glucose Test Tolerance (OGTT) after consumption of a high sugar load.
Evaluation of transcriptome analysis. | after 28 days of treatment
  Profile Evaluation of leukocyte gene expression through nutrigenomics study after consumption capsules containing standardized amount of yerba mate. The genes involved in lipid metabolism are isolated, identified and quantitated by real-time PCR technique. The results are expressed according to the identification and the number of genes.

SECONDARY OUTCOMES:
Clinical evaluation: arterial pressure (mean of three measurements for each 5 minutes). | 28 days
Clinical evaluation: waist circumference. | 28 days
Clinical evaluation: pulse. | 28 days
Clinical evaluation: weight. | 28 days
  weight in kg

CONTACTS AND LOCATIONS:
Overall Officials: Karimi S Gebara, MSc, Study Chair — Universidade Federal da Grande Dourados; Euclides L Cardozo Júnior, PhD, Principal Investigator — Universidade Paranaense
Locations (1):
- Euclides Lara Cardozo Júnior, Toledo, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Filip R, Lopez P, Giberti G, Coussio J, Ferraro G. Phenolic compounds in seven South American Ilex species. Fitoterapia. 2001 Nov;72(7):774-8. doi: 10.1016/s0367-326x(01)00331-8. PMID 11677016
- [Background] Alikaridis F. Natural constituents of Ilex species. J Ethnopharmacol. 1987 Jul;20(2):121-44. doi: 10.1016/0378-8741(87)90084-5. PMID 3657245
- [Background] Cardozo EL Jr, Cardozo-Filho L, Filho OF, Zanoelo EF. Selective liquid CO2 extraction of purine alkaloids in different Ilex paraguariensis progenies grown under environmental influences. J Agric Food Chem. 2007 Aug 22;55(17):6835-41. doi: 10.1021/jf0706225. Epub 2007 Jul 25. PMID 17650001
- [Background] Ghosh D, Scheepens A. Vascular action of polyphenols. Mol Nutr Food Res. 2009 Mar;53(3):322-31. doi: 10.1002/mnfr.200800182. PMID 19051188
- [Background] Cardozo Junior EL, Morand C. Interest of Mate (Ilex paraguariensis A.St.-Hil.) as a new natural functional food to preserve human cardiovascular health - A review. Journal of Functional Foods 21: 440-454, 2016.
- [Result] Arts IC, Hollman PC. Polyphenols and disease risk in epidemiologic studies. Am J Clin Nutr. 2005 Jan;81(1 Suppl):317S-325S. doi: 10.1093/ajcn/81.1.317S. PMID 15640497
- [Result] Balzan S, Hernandes A, Reichert CL, Donaduzzi C, Pires VA, Gasparotto A Jr, Cardozo EL Jr. Lipid-lowering effects of standardized extracts of Ilex paraguariensis in high-fat-diet rats. Fitoterapia. 2013 Apr;86:115-22. doi: 10.1016/j.fitote.2013.02.008. Epub 2013 Feb 17. PMID 23422228
- [Result] Chanet A, Milenkovic D, Deval C, Potier M, Constans J, Mazur A, Bennetau-Pelissero C, Morand C, Berard AM. Naringin, the major grapefruit flavonoid, specifically affects atherosclerosis development in diet-induced hypercholesterolemia in mice. J Nutr Biochem. 2012 May;23(5):469-77. doi: 10.1016/j.jnutbio.2011.02.001. Epub 2011 Jun 17. PMID 21684135
- [Result] Hooper L, Kroon PA, Rimm EB, Cohn JS, Harvey I, Le Cornu KA, Ryder JJ, Hall WL, Cassidy A. Flavonoids, flavonoid-rich foods, and cardiovascular risk: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2008 Jul;88(1):38-50. doi: 10.1093/ajcn/88.1.38. PMID 18614722